CLINICAL TRIAL: NCT05765916
Title: An Online Psychosocial Intervention for Fear of Cancer Recurrence in Breast Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, LYU Mengmeng, Principal Investigator, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LMengmeng
Record Dates: First submitted 2022-10-11; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Fear of Cancer Recurrence; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a two-armed RCT with a 1:1 allocation ratio: (1) an online mindfulness and acceptance therapy-based intervention; and (2) treat as usual.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online mindfulness and acceptance intervention (Experimental): Participants of the intervention group will receive an intervention manual and videos. The duration of the intervention will be six weeks. Participants will be asked for a minimum time investment of 60 min per week. The intervention will be delivered via WeChat video call. The intervention will be conducted following the intervention manual to ensure consistency of intervention content that delivered.
  Interventions: Behavioral: Online mindfulness and acceptance intervention
- Standard of care (No Intervention): Participants of the control group will be received usual follow-up care including regular medical checkups, which may include a physical exam, blood tests, and imaging tests.

INTERVENTIONS:
Behavioral: Online mindfulness and acceptance intervention — Session 1 aims to encourage participants to share their experiences; and introduce the purpose, content, delivery mode, duration, and frequency of the intervention.
  Session 2 aims to explain how negative illness perceptions lead to fear of cancer recurrence; and introduce the signs, screening, treatment and prognosis of breast cancer, ways to reduce the risk of recurrence, and symptom management.
  Session 3 aims to guide the participants to practice body scan and seated meditation.
  Session 4 aims to guide the participants to practice detached mindfulness, promoting reflection on the negative effect of indulging in unhelpful thoughts.
  In session 5, participants will receive several forms covering work, health, parenting style, intimate relationships, self-development and so on. Participant will be asked to choose one or two forms and set action plans.
  In session 6, the facilitator will invite participants to recall positive experiences and practice the "Self-care" exercise.
  Arms: Online mindfulness and acceptance intervention

SUMMARY:
A total of 244 breast cancer survivors will be invited to participate in the randomized controlled trial. Breast cancer survivors who meet the inclusion criteria and provide digital informed consent will be included. Participants will be stratified and randomized by the severity of baseline fear of cancer recurrence and time since diagnosis. In the control arm, women will be treated as usual. In the intervention arm, women will be offered a six-weekly, 60 min, online mindfulness and acceptance intervention. An online questionnaire will be used to collect data at four time points: before the first group session, immediately after the intervention, three months, and six months post-intervention. Phone interviews exploring participants' experiences will be held immediately after the intervention with women of the intervention group.

DETAILED DESCRIPTION:
The main study is a two-armed RCT with a 1:1 allocation ratio: (1) online psychosocial intervention; and (2) treat as usual. RCT is a gold standard for examining intervention effectiveness as it is the most reliable approach for proving the causal relationships between interventions and changes in outcome variables. Although no separate study can prove causality, randomization can reduce allocation bias stemmed from the differences in baseline variables and provides a rigorous approach for examining causality between interventions and outcome changes. Therefore, this study adopted an RCT design to examine the effectiveness of the psychosocial intervention in reducing FCR. Primary and secondary outcomes were assessed at two time points: before intervention commencement (T0) and immediate post-intervention (T1). Participants' experience in participating in the intervention was explored at the T1 through individual interview via phone call.

The magnitude of the effects of the intervention on the primary outcome of FCR and other secondary outcomes will be examined to determine if they were consistent with the existing literature. This study hypothesizes that the online psycho-social intervention will yield larger reductions in FCR and other psychosocial outcomes at post-treatment compared with a standardized care control group receiving formal follow-up care including clinical examination and health education on side-effects managements.

Research questions

Question 1: Primary outcome Is the online mindfulness and acceptance intervention effective in the reduction of FCR compared with control condition at post-intervention?

Question 2: Secondary outcomes Is the online mindfulness and acceptance intervention effective in reducing cognitive avoidance, illness representation, and in enhancing quality of life compared with the control condition?

Question 3: Participants' Experience What is the perception of the participants about the impact of the online intervention program on FCR?

ELIGIBILITY:
Inclusion Criteria:

* are over 18 years old
* diagnosed with primary stage 0-III breast cancer
* have completed primary cancer treatment within ten years (ongoing endocrine therapy is permitted)
* have sub-clinical or clinical fear of cancer recurrence as defined by a score in the range of 13 to 21 or > 21 on the fear of cancer recurrence inventory (FCRI)
* have a smart-phone
* can speak and read Mandarin

Exclusion Criteria:

* with cognitive impairment such as diagnosis of Parkinson's disease
* have clinically diagnosed psychiatric disorder
* are engaging in mindfulness and acceptance intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Fear of cancer recurrence | Change from the baseline FCRI score at six weeks.
  The Fear of Cancer Recurrence Inventory (FCRI) is a multidimensional self-reported instrument that assesses participants' experiences of FCR. The FCRI comprises 42 items and seven sub-scales inclusive of triggers, severity, psychological distress, functional impairment, insight, reassurance, and coping strategies. Responses are based on a 5-point Likert scale ranging from 0 (not at all or never) to 4 (a great deal or all the time). A total score can be obtained for each subscale and for the total scale by summing the items. The severity subscale is used to assess the severity of FCR. The sum of the items of severity subscale ranges from 0 to 36. Cut-offs for the severity subscale scores are as follows: nonclinical FCR, less than 13; subclinical FCR, 13 to 21; and clinically significant FCR, more than 21. The reliability and validity of the Chinese version of FCRI have been examined in 297 Chinese BCSs (Cronbach's alpha = 0.912; test-retest reliability = 0.88).

SECONDARY OUTCOMES:
Illness representation | Change from the baseline score of BIPQ-R at six weeks.
  Brief Illness Perception Questionnaire-Revised (BIPQ-R) is a nine-item self-reported instrument. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7). Responses are based on a 10-point Likert scale ranging from 0 (no at all) to 10 (extremely concerned). A total score can be obtained for each subscale and for the total scale by summing the items, with higher scores indicating more negative illness perceptions. Causal representations were assessed with an open-ended response item adapted from the IPQ-R that asked patients to list the three most important causal factors in their disease (item 9). The Cronbach's alpha values of the scale was 0.77 and the split-half reliability was 0.81.
Cognitive avoidance | Change from the baseline score of cognitive avoidance at six weeks.
  The Impact of Event Scale (IES) is a self-administered questionnaire that designed to tap into the two most common patterns of psychological reactions associated with trauma, namely intrusiveness (individuals involuntarily has those images, thoughts, nightmares, and feelings about the traumatic events) and avoidance (individuals intentionally do not want to think or talk about the traumatic event and all matters related to it). Weiss and Marmar added six items to the IES that measured emotional arousal - certain intrusive images and thoughts that provoke anxiety and worry - to develop a 22-item IES-R. Each item was measured using 5-point Likert scales, with higher mean scores on each subscale indicate greater avoidance/intrusiveness/arousal. In this study only avoidance subscale was used. The Chinese version IES-R subscales have good internal consistency (Cronbach's α = .83-.89).
Physical, role, emotional, social and cognitive functioning | Change from the baseline physical, role, emotional, social and cognitive functioning at six weeks.
  The European Organization for Research and Treatment-QOL breast cancer specific module (EORTC QOL-BR23): The 23-item EORTC QLQ-BR23 is composed of 5 dimensions to evaluate systemic therapy side effects, arm symptoms, breast symptoms, body image, and sexual functioning; 3 independent items assess sexual enjoyment, feeling of upset due to hair loss, and future perspective. These 23 items are rated on a 4-point Likert scale ranging from 1 (not at all) to 4 (very much). Responses are based on the frequency of cancer-related symptoms or distress an individual has experienced in the past week. The initial scale has demonstrated acceptable to good internal consistency (Cronbach's alpha = 0.52 to 0.89) and moderate to strong test-retest reliability (Pearson correlations ranging from 0.54 to 0.63). The reliability of the Chinese version of the EORTC QLQ-BR53 has been examined in Chinese cancer patients (Cronbach's alpha = 0.615 to 0.923).

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Chiew-Jiat SIAH, Dr, Study Director — National University of Singapore; Karis Kin Fong CHENG, Study Director — Global Nursing Research Center, Graduate School of Medicine, The University of Tokyo, Japan
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No